CLINICAL TRIAL: NCT06968611
Title: Improving Patient-centered Care for Diabetes in Bangladesh Through "Dynamic Integration" of Vision Care on the Demand Side
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orbis (Other)
Collaborators: District Diabetes Hospital, Dinajpur district of Bangladesh (Unknown); Gausul Azam BNSB Eye Hospital, Dinajpur district of Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PIS-DR-DEMAND-2025
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy (DR)
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Automated voice message exam reminder only (No Intervention): Participants will only receive an automated voice message reminder about the date of exam
- Intervention Group: Automated voice message + vision education + free reading glasses at appointment (Experimental): Participants will receive an automated voice message reminder about the date of the exam. Additionally, the participant will receive a message underscoring the risk of vision loss from poorly controlled DM, stressing that excellent compliance with visits and medications nearly completely eliminates this risk, and the participant will receive a free pair of reading glasses on first appointment.
  Interventions: Other: Education/information of risk; Other: Free eye glasses

INTERVENTIONS:
Other: Education/information of risk — Participant will receive a message underscoring risk of vision loss from poorly controlled DM, and how this risk can be largely eliminated with excellent compliance with mediations and clinical visits.
  Arms: Intervention Group: Automated voice message + vision education + free reading glasses at appointment
Other: Free eye glasses — Participants will receive a free pair of reading glass at their first appointment
  Arms: Intervention Group: Automated voice message + vision education + free reading glasses at appointment

SUMMARY:
The goal of this clinical trial is to determine whether there is an increase in participant uptake of diabetes mellitus (DM) and diabetic retinopathy (DR) services and improved quality of patient-centered diabetic care resulting from the use of automated voice message reminders to sensitize people with DM about the potential for sight loss alongside the provision of free reading glasses.

The main questions it aims to answer are:

1. Will the proportion of patients completing their scheduled DR and DM appointments within 3 weeks of the scheduled date be significantly increased in the group receiving the automated voice messages containing both appointment reminders and messaging about the importance of visit and medication compliance in reducing the risk of vision loss, compared with participant messages which only remind them of their appointments?
2. What is the cost-effectiveness, measured as total intervention cost per additional patient complying with the suggested exam?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DM within the last 6 months
* Over 30 years of age
* Currently treated at the Dinajpur Diabetes Hospital
* Possess a mobile phone to receive voice messages
* Willingness to participate in the study, and ability to give informed consent

Exclusion Criteria:

* Other significant causes of vision loss
* Medical conditions that could impair compliance with follow-up (such as stroke, dementia, etc.)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing their diabetes or DR exam within 3 weeks of the scheduled date. | 3 weeks following scheduled exam date

SECONDARY OUTCOMES:
Cost-effectiveness, measured as total intervention cost per additional patient adherence with the suggested exam. | Enrollment to 3 weeks following suggested exam date

CONTACTS AND LOCATIONS:
Overall Officials: Munir Ahmed, Principal Investigator — Orbis Bangladesh; Nathan Congdon, Principal Investigator — Orbis
Locations (2):
- Bangladesh (2):
  - Gausul Azam BNSB Eye Hospital, Dinajpur
  - Dinajpur Diabetes & Swasthoseba Hospital, Dinajpur Sadar

IPD SHARING:
Plan to Share IPD: Yes
de-identified data is available upon reasonable request to the corresponding author following the study completion
Supporting Information: Study Protocol, SAP, ICF